CLINICAL TRIAL: NCT01581827
Title: SCREEN-HFL (SCReening Evaluation of the Evolution of New Heart Failure) - a Longitudinal Study
Acronym: SHF-L
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Senior Lecturer, Monash University
Other Study IDs: 52/09
Record Dates: First submitted 2012-04-12; First posted 2012-04-20 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; BNP; NT-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to measure BNP and NT-proBNP
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: People at high risk of heart failure (from SCREEN-HF study)

SUMMARY:
Heart failure (when the heart does not pump as well as it used to) is a medical condition which reduces the quality of life for the sufferers. Approximately 10% of people in western societies aged over 75 develop heart failure. There has been a shift towards prevention of this disease and it is hoped that BNP (brain natriuretic peptides) and NT-proBNP (N-terminal proBNP) will prove to be useful indicators of those at greatest risk. The current study therefore plans to follow up the 3500 participants at risk of heart failure from the original SCREEN-HF study.

Participants who are willing to participate will be contacted annually. They will undergo a short physical exam, will be asked to complete a Quality of Life questionnaire and will have a blood sample taken. At the end of the study participants will also have an ECG and an echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

1. Consented and enrolled in the SCREEN-HF study and who agreed to further contact
2. Age ≥ 60 years
3. Subjects at high-risk of subsequent development of heart failure; comprising at least one of:

   * Prior myocardial infarction (MI) without known left ventricular (LV) dysfunction
   * Current active ischaemic heart disease
   * Prior Cerebrovascular Accident (CVA)
   * Known valvular heart disease without known LV dysfunction
   * Atrial fibrillation
   * Treated hypertension, of at least 2 years duration
   * Treated Diabetes mellitus, of at least 2 years duration
   * Chronic renal impairment (eGFR < 60 ml/min)

Exclusion Criteria:

1. Known systolic or diastolic heart failure
2. LV systolic or diastolic dysfunction on echocardiography or other objective imaging modality (if known).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People at high risk of heart failure
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in NT-proBNP | baseline and 5 years
Change in echocardiogram | baseline and 5 years

SECONDARY OUTCOMES:
incidence of new heart failure | baseline and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University/Alfred Hospital
Locations (1):
- Monash University, Caulfield, Victoria, Australia

REFERENCES:
- [Derived] Campbell DJ, Coller JM, Gong FF, McGrady M, Boffa U, Shiel L, Liew D, Stewart S, Owen AJ, Krum H, Reid CM, Prior DL. Kidney age - chronological age difference (KCD) score provides an age-adapted measure of kidney function. BMC Nephrol. 2021 Apr 26;22(1):152. doi: 10.1186/s12882-021-02324-y. PMID 33902478
- [Derived] Gong FF, Jelinek MV, Castro JM, Coller JM, McGrady M, Boffa U, Shiel L, Liew D, Wolfe R, Stewart S, Owen AJ, Krum H, Reid CM, Prior DL, Campbell DJ. Risk factors for incident heart failure with preserved or reduced ejection fraction, and valvular heart failure, in a community-based cohort. Open Heart. 2018 Jul 23;5(2):e000782. doi: 10.1136/openhrt-2018-000782. eCollection 2018. PMID 30057766